CLINICAL TRIAL: NCT02789891
Title: Randomized Controlled Trials on Laparoscopic No. 14v Lymph Node Dissection for Advanced Lower Third Gastric Cancer
Brief Title: Randomized Controlled Trials on Laparoscopic No. 14v LNS Dissection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Director, Principal Investigator, Clinical Professor, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-03
Record Dates: First submitted 2016-05-29; First posted 2016-06-03 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- D2 Lymphadenectomy including No. 14v (Experimental): Laparoscopic distal gastrectomy with D2 lymphadenectomy including No. 14v lymph node dissection will be performed for the treatment of patients assigned to this group
  Interventions: Procedure: D2 lymphadenectomy including No. 14v
- D2 lymphadenectomy excluding No. 14v (Active Comparator): Laparoscopic distal gastrectomy with D2 lymphadenectomy excluding No. 14v lymph node dissection will be performed for the treatment of patients assigned to this group
  Interventions: Procedure: lymphadenectomy excluding No. 14v

INTERVENTIONS:
Procedure: D2 lymphadenectomy including No. 14v — After exclusion of T4b, or distant metastasis case by diagnostic laparoscopy, Laparoscopic distal with D2 lymphadenectomy including No. 14v Lymph Node Dissection will be performed with curative treated intent. The type of reconstruction will be selected according to the surgeon's experience
  Arms: D2 Lymphadenectomy including No. 14v
Procedure: lymphadenectomy excluding No. 14v — After exclusion of T4b, or distant metastasis case by diagnostic laparoscopy, Laparoscopic distal gastrectomy with D2 lymphadenectomy excluding No. 14v Lymph Node Dissection will be performed with curative treated intent. The type of reconstruction will be selected according to the surgeon's experience
  Arms: D2 lymphadenectomy excluding No. 14v

SUMMARY:
The purpose of this study is to explore the short-term, long-term and oncological outcomes of laparoscopic No. 14v lymph node dissection in advanced lower third gastric cancer.

DETAILED DESCRIPTION:
A prospective randomized comparison of laparoscopic No. 14v lymph node dissection in advanced lower third gastric cancer will be performed, to evaluate the short-term, long-term and oncological outcomes. The evaluation parameters are perioperative clinical efficacy, postoperative life quality, immune function and 3-year survival and recurrence rates.

ELIGIBILITY:
Inclusion Criteria:• Age from 18 to 75 years

* Primary lower third gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
* cT2-4a, N0-3, M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual Seventh Edition
* No distant metastasis is observed. And the spleen, pancreas or other adjacent organs are not involved by the tumor.
* Performance status of 0 or 1 on Eastern Cooperative Oncology Group scale (ECOG)
* American Society of Anesthesiology score (ASA) class I, II, or III
* Written informed consent

Exclusion Criteria:• Women during pregnancy or breast-feeding

* Severe mental disorder
* History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
* History of previous gastrectomy, endoscopic mucosal resection or endoscopic submucosal dissection
* Enlarged or bulky regional lymph node envelop important vessels
* History of other malignant disease within past five years
* History of previous neoadjuvant chemotherapy or radiotherapy
* History of unstable angina or myocardial infarction within past six months
* History of cerebrovascular accident within past six months
* History of continuous systematic administration of corticosteroids within one month
* Requirement of simultaneous surgery for other disease
* Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
* FEV1<50% of predicted values

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
3-year disease overall survival rate | 36 months

SECONDARY OUTCOMES:
No.14v Lymph node metastasis rate | 10 days
Morbidity and mortality | 30 days; 36 months
  The early postoperative complication and mortality are defined as the event observed within 30 days after surgery, while the time frame for late complication is the period from postoperative day 31th to the end of month 36th.
3-year free survival rate | 36 months
3-year recurrence pattern | 36 months
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type
Time to first ambulation | 10 days
  The data of postoperative recovery course.
The number of lymph node dissection | 10day
The variation of weight | 12 months
  The variation of weight on postoperative 3, 6, 9 and 12 months
The daily highest body temperature | 7 day
  The daily highest body temperature before discharge
Time to first flatus | 10 days
Time to first liquid diet | 10 days
Time to soft diet | 10 days
Duration of hospital stay | 10 days
The amount of abdominal drainage | 10 days
Blood transfusion | 10 days
The number of positive lymph nodes | 1 day
Intraoperative lymph node dissection time | 1 day
  intraoperative No.14v lymph node dissection time includes infrapyloric area lymph node,suprapancreatic area lymph node,splenic hilar area lymph node, cardial area lymph node
Intraoperative blood loss | 1 day
Intraoperative injury | 1 day
The amount of use of titanium clip | 1 day
The rate of conversion to laparotomy | 1 day
The variation of cholesterol | 12 months
  The variation of cholesterol on postoperative 3, 6, 9 and 12 months
The variation of albumin | 12 months
  The variation of albumin on postoperative 3, 6, 9 and 12 months
The results of endoscopy | 12 months
  the results of endoscopy on postoperative 3 and 12 months
The values of white blood cell count | 7 days
  the values of white blood cell count from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded
The values of hemoglobin | 7 days
  and the values of hemoglobin from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded.
The values of C-reactive protein | 7 days
  and the values of C-reactive protein from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded.
The values of prealbumin | 7 days
  and the values of prealbumin from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded.
The values of relevant immune cytokines | 7 days
  and the values of relevant immune cytokines including T cell percentage, T-helper lymphocytes (CD4+) percentage, T-suppressor lymphocytes (CD8+) percentage, natural killer (NK) cells percentage from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded.
Visual Analog Score for pain | 7 days
  the values of visual analog score for pain before operation and on postoperative day 1 to day 7 are recorded.
EORTC QLQ-C30 and QLQ - STO22 | Time Frame: 36 months
  European Organization fo Research and Treatment(EORTC) QLQ-C30 and QLQ - STO22 before operation and on postoperative month 6,12,36 are recorded.